CLINICAL TRIAL: NCT03925402
Title: Ertapenem for Initial Empirical Treatment of Third Generation Cephalosporin Resistant Enterobacteriaceae Bacteremia: a Propensity Score Analysis
Brief Title: Ertapenem for Initial Empirical Treatment of Third Generation Cephalosporin Resistant Enterobacteriaceae Bacteremia
Status: Completed | Type: Observational
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AMED2019
Record Dates: First submitted 2019-04-20; First posted 2019-04-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Bacteremia; Infection, Bacterial
MeSH Terms: conditions — Bacteremia; Bacterial Infections | interventions — Ertapenem; Carbapenems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ertapenem: Patients who received ertapenem as an empirical antibiotic
  Interventions: Drug: Ertapenem
- Other carbapenems: Patients who received carbapenems other than ertapenem as an empirical antibiotic
  Interventions: Drug: Carbapenems

INTERVENTIONS:
Drug: Ertapenem — Ertapenem injection
  Groups: Ertapenem
Drug: Carbapenems — Other carbapenems injection
  Groups: Other carbapenems

SUMMARY:
This study aims to assess whether ertapenem as an empiric treatment of third-generation-cephalosporin resistant Enterobacteriaceae (3GCRE) bacteremia is non-inferior to other carbapenems in term of 30-day mortality.

DETAILED DESCRIPTION:
There are limited data of the efficacy of ertapenem as the empiric treatment of serious invasive infections, such as bloodstream infections (BSIs), that are due to ESBL-producing Enterobacteriaceae. Previous studies of ertapenem were done in small group of patients, in less invasive infection, as a definite 'step-down' therapy, or as compared to other non-carbapenem antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Adults, either sex, ages 18 years or above
* Patients with 3GCRE bacteremia
* Patients admitted to any of the study sites

Exclusion Criteria:

* Discontinuation of antibiotic due to transition to hospice care
* Polymicrobial bacteremia
* Empirical antibiotic after 24 hours of first evidence of bacteremia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older admitted to Phramongkutklao Hospital, and Ananda Mahidol Hospital with 3GCRE monomicrobial bacteremia will be prospectively identified. In given a patient, only the initial episode of 3GCRE monomicrobial bacteremia during the study period will be included.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  death from any cause within 30 days after the blood culture with bacteraemia is drawn

SECONDARY OUTCOMES:
In-hospital mortality | 90 days
  death from any cause within the duration of admission with bacteraemia
14-day mortality | 14 days
  death from any cause within 14 days after the blood culture with bacteraemia is drawn
90-day mortality | 90 days
  death from any cause within 90 days after the blood culture with bacteraemia is drawn
• Length of stay | 90 days
  Duration of admission with bacteraemia

CONTACTS AND LOCATIONS:
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasikasin V, Panuvatvanich B, Rawson TM, Holmes AH, Nasomsong W. Towards optimizing carbapenem selection in stewardship strategies: a prospective propensity score-matched study of ertapenem versus class 2 carbapenems for empirical treatment of third-generation cephalosporin-resistant Enterobacterales bacteraemia. J Antimicrob Chemother. 2023 Jul 5;78(7):1748-1756. doi: 10.1093/jac/dkad165. PMID 37252945